CLINICAL TRIAL: NCT02725749
Title: Effect of Low Level Laser Therapy Associated With Exercise in Subacromial Impingement Syndrome: a Randomized, Double-blind Study
Brief Title: Low Level Laser Therapy Associated With Exercise in Subacromial Impingement Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Raquel A. Casarotto, PHD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USaoPauloGH1
Record Dates: First submitted 2016-03-21; First posted 2016-04-01 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Subacromial Impingement Syndrome
Keywords: shoulder; low level laser therapy; exercises
MeSH Terms: conditions — Shoulder Impingement Syndrome; Motor Activity | interventions — Lasers; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Laser (Experimental)
  Interventions: Radiation: Laser
- Exercise (Experimental)
  Interventions: Other: EXE
- Laser and Exercise (Experimental)
  Interventions: Radiation: Laser + EXE

INTERVENTIONS:
Radiation: Laser — Laser used were GaAs (904 nm, 60 mW), in continuous emission. The participants received application of laser three times or week for eight weeks, on 9 shoulder points (3 Joules/point) per session.
  Arms: Laser
Other: EXE — Isotonic strengthening exercises were performed for the scapular pivot, scapula stabilizer, and humeral propellant muscle groups. Three sets of 15 repetitions of each isotonic strengthening exercise were performed. The isometric exercises were performed in ten sets of ten seconds each. Analytical stretching of each muscle group was performed at the beginning of the session for 30 seconds.
  The participants performed the exercises three times a week for eight weeks.
  Other Names: Exercise
  Arms: Exercise
Radiation: Laser + EXE — Laser used were GaAs (904 nm, 60 mW), in continuous emission. The participants received application of laser three times or week for eight weeks, on 9 shoulder points (3 Joules/point) per session.
  Isotonic strengthening exercises were performed for the scapular pivot, scapula stabilizer, and humeral propellant muscle groups. Three sets of 15 repetitions of each isotonic strengthening exercise were performed. The isometric exercises were performed in ten sets of ten seconds each. Analytical stretching of each muscle group was performed at the beginning of the session for 30 seconds.
  The participants performed the exercises three times a week for eight weeks.
  Other Names: Laser and Exercise
  Arms: Laser and Exercise

SUMMARY:
Objectives: The objective was to compare low level laser therapy (LLLT) therapy versus low LLLT therapy in combination with an exercise or exercise only on pain, range of motion (ROM), functionality, and activity limitation in patients with subacromial impact syndrome.

Design: Randomized and placebo-controlled clinical trial.

Setting: The setting for the study was the Municipal Clinic of Barueri, São Paulo, Brazil.

Participants: 60 patients with subacromial impact syndrome were randomly assigned in three groups.

Interventions: Group I, experimental (n=21) treated with low level laser therapy and exercises; Group II, experimental (n=21) treated with exercises; and Group III, experimental (n=18) treated with low level laser therapy. Laser used were GaAs (904 nm, 60 mW), in continuous emission. The participants received application of laser three times or week for eight weeks, on 9 shoulder points (3 Joules/point) per session.

Main outcome measures: Visual Analogic Scale (VAS) score, Shoulder Pain and Disability Index (SPADI), goniometer, Modified-University of California at Los Angeles Shoulder Rating Scale (UCLA), recorded before and after treatment.

DETAILED DESCRIPTION:
In the groups that received low level laser therapy (LLLT), energy was irradiated over three insertion points in the supraspinatus muscle region, three points on the bursa subacromial, and three points along the bicipital groove, at 3 Joules per point. Total dose per shoulder was 27 Joules per treatment, using a previously calibrated Irradia Class 3B (Stockholm, Sweden). Pen's semiconductor consisted of gallium arsenide with a wavelength of 904 nm, frequency of 700 Hz, average potency of 60 mW, peak potency of 20 W, pulse duration of 4.3 ms, and 50 seconds per point (0.5cm2 area). The parameters followed the recommendation of the World Association of Laser Therapy for subacromial impact syndrome.

The participants received application of laser three times or week for eight weeks.

The groups treated with exercise followed the same training program. Isotonic strengthening exercises were performed for the scapular pivot, scapula stabilizer, and humeral propellant muscle groups. Three sets of 15 repetitions of each isotonic strengthening exercise were performed. The isometric exercises were performed in ten sets of ten seconds each. Analytical stretching of each muscle group was performed at the beginning of the session for 30 seconds.

The participants performed the exercises three times a week for eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of subacromial impact syndrome
* Age range: 30-75 years
* Both genders

Exclusion Criteria:

* cancer,
* diabetes,
* symptomatic shoulder osteoarthritis,
* surgery or previous fractures in the humeral head of the shoulder,
* history of acute trauma, calcification of the articular rotator tendon,
* total tendon rupture,
* cervical myofascial syndrome,
* radicular pain,
* inflammatory rheumatic disease,
* neurological disorders,
* depressive syndrome
* use of antidepressants,
* use of anti-inflammatory medications
* use anxiolytics

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pain assessed using a VAS | 1 year
  Pain was assessed using a VAS consisting of a 10cm ruler (without numbers), ranging from "no pain" on the left side to "unbearable pain" on the right side. The patients were instructed to mark their level of pain on the ruler.
Range of motion assessed with a universal goniometer (Aesculap) | 1 year
  Range of motion was assessed with a universal goniometer (Aesculap) used to measure shoulder flexion and extension according to the methods described by Marques et al. (2011).
Functionality measured using the Modified-University of California at Los Angeles Shoulder Rating Scale | 1 year
  Functionality was measured using the Modified-University of California at Los Angeles Shoulder Rating Scale, which consists of five domains-pain, function, range of motion, muscle strength, and patient satisfaction-and a possible total of 35 points, with higher scores indicating better results
Quality of life assessed with the Shoulder Pain and Disability Index (SPADI) | 1 year
  Quality of life was assessed with the Shoulder Pain and Disability Index (SPADI). This questionnaire, which is specific to the shoulder joint, assesses pain and disability. The SPADI consists of 13 items distributed in the areas of pain (five items) and function (eight items), with each item scored on a numerical scale from 0 to 10 points. The final score of the questionnaire and the score of each domain are converted into percentages ranging from 0 to 100%, with higher scores indicating worse shoulder conditions

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alfredo PP, Bjordal JM, Junior WS, Marques AP, Casarotto RA. Efficacy of low-level laser therapy combined with exercise for subacromial impingement syndrome: A randomised controlled trial. Clin Rehabil. 2021 Jun;35(6):851-860. doi: 10.1177/0269215520980984. Epub 2020 Dec 14. PMID 33307783